CLINICAL TRIAL: NCT04827134
Title: A Randomized, 2-Cohort, 2-Period, Single Dose, Crossover Clinical Study to Assess the Effect of Food on the Pediatric Dispersible Tablet Formulations of TRIUMEQ (Dolutegravir/Abacavir/Lamivudine) and DOVATO (Dolutegravir/Lamivudine) in Healthy Adult Participants
Brief Title: A Food-effect Study of the Pediatric Dispersible Tablet Formulations of TRIUMEQ® and DOVATO® in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 216149
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2022-06

CONDITIONS: HIV Infections
Keywords: TRIUMEQ; DOVATO; Pharmacokinetics; Food effect; Dolutegravir; Abacavir; Lamivudine
MeSH Terms: conditions — HIV Infections | interventions — abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-dose, 2-cohort, 2-period crossover study.
Masking Description: This is an open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: TRIUMEQ Fed followed by TRIUMEQ Fasted (Experimental): Participants received TRIUMEQ (dolutegravir [DTG] 5 milligram [mg]/abacavir [ABC] 60 mg/lamivudine [3TC] 30 mg), dispersible tablets administered as a dispersion immediately after a high calorie meal (under fed condition) (Treatment A) in treatment period 1 followed by TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg), dispersible tablets administered as a dispersion under fasted conditions (Treatment B) in treatment period 2. The treatment periods were separated by a washout period of about 7 days. All participants were followed-up for 7 to 14 days of last dose in treatment period 2.
  Interventions: Drug: TRIUMEQ
- Cohort 1: TRIUMEQ Fasted followed by TRIUMEQ Fed (Experimental): Participants received TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg), dispersible tablets administered as a dispersion under fasted conditions (Treatment B) in treatment period 1 followed by TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg), dispersible tablets administered as a dispersion immediately after a high calorie meal (under fed condition) (Treatment A) in treatment period 2. The treatment periods were separated by a washout period of about 7 days. All participants were followed-up for 7 to 14 days of last dose in treatment period 2.
  Interventions: Drug: TRIUMEQ
- Cohort 2: DOVATO Fed followed by DOVATO Fasted (Experimental): Participants received DOVATO (DTG 5 mg/3TC 30 mg), dispersible tablets administered as a dispersion immediately after a high calorie meal (under fed condition) (Treatment C) in treatment period 1 followed by DOVATO (DTG 5 mg/3TC 30 mg), dispersible tablets administered as a dispersion under fasted conditions (Treatment D) in treatment period 2. The treatment periods were separated by a washout period of about 7 days. All participants were followed-up for 7 to 14 days of last dose in treatment period 2.
  Interventions: Drug: DOVATO
- Cohort 2: DOVATO Fasted followed by DOVATO Fed (Experimental): Participants received DOVATO (DTG 5 mg/3TC 30 mg), dispersible tablets administered as a dispersion under fasted conditions (Treatment D) in treatment period 1 followed by DOVATO (DTG 5 mg/3TC 30 mg), dispersible tablets administered as a dispersion immediately after a high calorie meal (under fed condition) (Treatment C) in treatment period 2. The treatment periods were separated by a washout period of about 7 days. All participants were followed-up for 7 to 14 days of last dose in treatment period 2.
  Interventions: Drug: DOVATO

INTERVENTIONS:
Drug: TRIUMEQ — TRIUMEQ will be available as fixed dose combination (FDC) dispersible tablets to be administered orally as a dispersion.
  Arms: Cohort 1: TRIUMEQ Fasted followed by TRIUMEQ Fed; Cohort 1: TRIUMEQ Fed followed by TRIUMEQ Fasted
Drug: DOVATO — DOVATO will be available as FDC dispersible tablets to be administered orally as a dispersion.
  Arms: Cohort 2: DOVATO Fasted followed by DOVATO Fed; Cohort 2: DOVATO Fed followed by DOVATO Fasted

SUMMARY:
This study will assess the effect of food on the pharmacokinetics (PK) of pediatric formulations of TRIUMEQ (dolutegravir [DTG] 5 milligrams [mg]/abacavir [ABC] 60 mg/lamivudine [3TC] 30 mg) dispersible tablets and DOVATO (DTG 5 mg/3TC 30 mg) dispersible tablets in healthy adult participants. Additionally, safety and tolerability of these formulations will also be assessed. TRIUMEQ and DOVATO are registered trademarks of GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and ECG).
* Body weight >=50.0 kilograms (kg) (110 pounds [lbs.]) for males and >=45 kg (99 lbs.) for females and body mass index within the range 18.5 to 31.0 kilogram per meter square (kg/m^2, inclusive).
* A male participant is eligible to participate if they agree to use contraceptive methods.
* A female participant is eligible to participate if she is not pregnant (, not lactating or breastfeeding, and at least 1 of the following conditions applies: Is not a woman of childbearing potential (WOCBP) OR Is a WOCBP and using a non-hormonal contraceptive method that is highly effective
* Capable of giving signed informed consent
* Documentation that the participant is negative for the human leukocyte antigen (HLA) B*5701 allele.

Exclusion Criteria:

* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Medical history of cardiac arrhythmias, prior myocardial infarction in the past 3 months, or cardiac disease or a family or personal history of long QT syndrome.
* A pre-existing condition interfering with normal gastrointestinal anatomy or motility (e.g., gastroesophageal reflux disease, gastric ulcers, gastritis), hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study intervention.
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 milliseconds (msec).
* A participant with known or suspected active coronavirus disease (COVID-19) infection OR contact with an individual with known COVID-19, within 14 days of study enrollment.
* Presence of hepatitis B surface antigen at screening or within 3 months prior to starting study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to starting study intervention AND positive on reflex to hepatitis C ribonucleic acid (RNA).
* Positive human immunodeficiency virus (HIV)-1 and -2 antigen/antibody immunoassay at screening.
* Alanine aminotransferase (ALT) >1.5 × upper limit of normal (ULN). A single repeat of ALT is allowed within a single screening period to determine eligibility.
* Bilirubin >1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat of any laboratory abnormality is allowed within a single screening period to determine eligibility.
* Any acute laboratory abnormality at screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Any Grade 2 to 4 laboratory abnormality at screening, with the exception of creatine phosphokinase (CPK) and lipid abnormalities (e.g., total cholesterol, triglycerides), and ALT (described above), will exclude a participant from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat of any laboratory abnormality is allowed within a single screening period to determine eligibility.
* A positive test result for drugs of abuse (including marijuana), alcohol, or cotinine (indicating active current smoking) at screening or before the first dose of study intervention.
* Unable to refrain from the use of prescription or non-prescription drugs including vitamins, herbal and dietary supplements (including St. John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study intervention and for the duration of the study until completion of the follow-up visit, unless, in the opinion of the investigator and ViiV Healthcare (VH)/GlaxoSmithKline medical monitor, the medication will not interfere with the study procedures or compromise participant safety.
* Unwillingness to abstain from excessive consumption of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos or their fruit juices within 7 days prior to the first dose of study intervention(s) until the end of the study.
* Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to Day 1 of Period 1 in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the study intervention (whichever is longer).
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within 60 days.
* Estimated serum creatinine clearance (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) <90 milliliter per minute (mL/min).
* History of regular alcohol consumption within 6 months of the study, defined as an average weekly intake of >14 units for males or >7 drinks for females.
* Unable to refrain from tobacco or nicotine-containing products within 1 month prior to screening.
* History of sensitivity, prior intolerance or hypersensitivity to any of the study interventions, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States.
Pre-assignment Details: A total of 33 participants (16 participants in Cohort 1 and 17 participants in Cohort 2) were enrolled in the study.
Period: Treatment Period 1 (1 Day)
Arm/Group | Cohort 1: TRIUMEQ Fed Followed by TRIUMEQ Fasted | Cohort 1: TRIUMEQ Fasted Followed by TRIUMEQ Fed | Cohort 2: DOVATO Fed Followed by DOVATO Fasted | Cohort 2: DOVATO Fasted Followed by DOVATO Fed
Started | 8 | 8 | 8 | 9
Completed | 8 | 8 | 7 | 9
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Washout Period (up to 7 Days)
Arm/Group | Cohort 1: TRIUMEQ Fed Followed by TRIUMEQ Fasted | Cohort 1: TRIUMEQ Fasted Followed by TRIUMEQ Fed | Cohort 2: DOVATO Fed Followed by DOVATO Fasted | Cohort 2: DOVATO Fasted Followed by DOVATO Fed
Started | 8 | 8 | 7 | 9
Completed | 8 | 8 | 7 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2 (1 Day)
Arm/Group | Cohort 1: TRIUMEQ Fed Followed by TRIUMEQ Fasted | Cohort 1: TRIUMEQ Fasted Followed by TRIUMEQ Fed | Cohort 2: DOVATO Fed Followed by DOVATO Fasted | Cohort 2: DOVATO Fasted Followed by DOVATO Fed
Started | 8 | 8 | 7 | 9
Completed | 8 | 8 | 7 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: TRIUMEQ Fed Followed by TRIUMEQ Fasted | Cohort 1: TRIUMEQ Fasted Followed by TRIUMEQ Fed | Cohort 2: DOVATO Fed Followed by DOVATO Fasted | Cohort 2: DOVATO Fasted Followed by DOVATO Fed | Total
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 33
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  19-64 years | 8 | 8 | 8 | 9 | 33
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 2 | 10
  Male | 6 | 4 | 6 | 7 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian: Central/South Asian Heritage | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 3 | 2 | 4 | 11
  White | 6 | 4 | 5 | 5 | 20
  Multiple: Black or African American & White | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero Extrapolated to Infinity (AUC [0-inf]) of DTG, ABC and 3TC Following Administration of TRIUMEQ Under Fed and Fasted Conditions
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of DTG, ABC and 3TC. The PK parameters were calculated by standard non-compartmental analysis
Time Frame: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 and 72 Hours post dose in each treatment periods 1 and 2
Population: Pharmacokinetic Parameter Population consisted of all participants who underwent plasma PK sampling and had evaluable (non-missing) PK parameters estimated. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed: Participants received TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg), dispersible tablets administered as a dispersion immediately after a high calorie meal (under fed condition) during Treatment Periods 1 and 2 of Cohort 1 of study
- Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted: Participants received TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg), dispersible tablets administered as a dispersion under fasted conditions during Treatment Periods 1 and 2 of Cohort 1 of study.
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Hours*nanogram per milliliter
  DTG | 59140 (25.7) | 67210 (24.0)
  ABC | 8565 (24.9) | 9986 (28.8)
  3TC: number analyzed (Participants) | 15 | 16
  3TC | 6508 (19.9) | 7295 (23.4)
Statistical Analysis 1: Comparison: Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed vs Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.8800, 90% CI 2-sided [0.8344 to 0.9282] — An analysis of variance (ANOVA) was performed on parameter AUC(0-inf) for Analyte DTG to compare treatment arms Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed with Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Statistical Analysis 2: Comparison: Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed vs Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.8578, 90% CI 2-sided [0.8168 to 0.9007] — An analysis of variance was performed on parameter AUC(0-inf) for Analyte ABC to compare treatment arms Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed with Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Statistical Analysis 3: Comparison: Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed vs Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.8919, 90% CI 2-sided [0.8316 to 0.9566] — An analysis of variance was performed on parameter AUC(0-inf) for Analyte 3TC to compare treatment arms Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed with Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted

2. Primary Outcome: Cohort 1: AUC From Time Zero to Time of Last Observed Quantifiable Concentration (AUC [0-t]) of DTG, ABC and 3TC Following Administration of TRIUMEQ Under Fed and Fasted Conditions
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of DTG, ABC and 3TC. The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Hours*nanogram per milliliter
  DTG | 55770 (23.8) | 63790 (22.7)
  ABC | 8501 (25.4) | 9923 (28.9)
  3TC | 6319 (18.9) | 7182 (23.5)
Statistical Analysis 1: Comparison: Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed vs Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.8744, 90% CI 2-sided [0.8293 to 0.9219] — An analysis of variance was performed on parameter AUC(0-t) for Analyte DTG to compare treatment arms Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed with Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Statistical Analysis 2: Comparison: Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed vs Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.8567, 90% CI 2-sided [0.8159 to 0.8995] — An analysis of variance was performed on parameter AUC(0-t) for Analyte ABC to compare treatment arms Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed with Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Statistical Analysis 3: Comparison: Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed vs Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.8798, 90% CI 2-sided [0.8202 to 0.9438] — An analysis of variance was performed on parameter AUC(0-t) for Analyte 3TC to compare treatment arms Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed with Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted

3. Primary Outcome: Cohort 1: Maximum Observed Concentration (Cmax) of DTG, ABC and 3TC Following Administration of TRIUMEQ Under Fed and Fasted Conditions
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Nanogram per milliliter
  DTG | 2359 (17.6) | 3322 (20.6)
  ABC | 1837 (21.1) | 4080 (32.3)
  3TC | 886.9 (18.9) | 1392 (33.3)
Statistical Analysis 1: Comparison: Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed vs Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.7102, 90% CI 2-sided [0.6598 to 0.7643] — An analysis of variance was performed on parameter Cmax for Analyte DTG to compare treatment arms Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed with Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Statistical Analysis 2: Comparison: Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed vs Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.4503, 90% CI 2-sided [0.3976 to 0.5100] — An analysis of variance was performed on parameter Cmax for Analyte ABC to compare treatment arms Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed with Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Statistical Analysis 3: Comparison: Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed vs Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.6373, 90% CI 2-sided [0.5594 to 0.7260] — An analysis of variance was performed on parameter Cmax for Analyte 3TC to compare treatment arms Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed with Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted

4. Primary Outcome: Cohort 2: AUC (0-inf) of DTG and 3TC Following Administration of DOVATO Under Fed and Fasted Conditions
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of DTG and 3TC. The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- Cohort 2: DOVATO (DTG/3TC) Fed: Participants received DOVATO (DTG 5 mg/3TC 30 mg), dispersible tablets administered as a dispersion immediately after a high calorie meal (under fed condition) during Treatment Periods 1 and 2 of Cohort 2 of study.
- Cohort 2: DOVATO (DTG/3TC) Fasted: Participants received DOVATO (DTG 5 mg/3TC 30 mg), dispersible tablets administered as a dispersion under fasted conditions during Treatment Periods 1 and 2 of Cohort 2 of study.
Arm/Group | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Hours*nanogram per milliliter
  DTG | 47830 (24.2) | 51800 (24.3)
  3TC | 6975 (10.1) | 7864 (13.9)
Statistical Analysis 1: Comparison: Cohort 2: DOVATO (DTG/3TC) Fed vs Cohort 2: DOVATO (DTG/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.9148, 90% CI 2-sided [0.8834 to 0.9472] — An analysis of variance was performed on parameter AUC(0-inf) for Analyte DTG to compare treatment arms Cohort 2: DOVATO (DTG/3TC) Fed with Cohort 2: DOVATO (DTG/3TC) Fasted
Statistical Analysis 2: Comparison: Cohort 2: DOVATO (DTG/3TC) Fed vs Cohort 2: DOVATO (DTG/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.8847, 90% CI 2-sided [0.8303 to 0.9426] — An analysis of variance was performed on parameter AUC(0-inf) for Analyte 3TC to compare treatment arms Cohort 2: DOVATO (DTG/3TC) Fed with Cohort 2: DOVATO (DTG/3TC) Fasted

5. Primary Outcome: Cohort 2: AUC (0-t) of DTG and 3TC Following Administration of DOVATO Under Fed and Fasted Conditions
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 17 | 16
Hours*nanogram per milliliter
  DTG | 46060 (22.2) | 49690 (22.0)
  3TC | 6799 (10.5) | 7762 (14.0)
Statistical Analysis 1: Comparison: Cohort 2: DOVATO (DTG/3TC) Fed vs Cohort 2: DOVATO (DTG/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.9163, 90% CI 2-sided [0.8862 to 0.9475] — An analysis of variance was performed on parameter AUC(0-t) for Analyte DTG to compare treatment arms Cohort 2: DOVATO (DTG/3TC) Fed with Cohort 2: DOVATO (DTG/3TC) Fasted
Statistical Analysis 2: Comparison: Cohort 2: DOVATO (DTG/3TC) Fed vs Cohort 2: DOVATO (DTG/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.8806, 90% CI 2-sided [0.8251 to 0.9398] — An analysis of variance was performed on parameter AUC(0-t) for Analyte 3TC to compare treatment arms Cohort 2: DOVATO (DTG/3TC) Fed with Cohort 2: DOVATO (DTG/3TC) Fasted

6. Primary Outcome: Cohort 2: Cmax of DTG and 3TC Following Administration of DOVATO Under Fed and Fasted Conditions
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 17 | 16
Nanogram per milliliter
  DTG | 2331 (15.4) | 3131 (19.8)
  3TC | 1084 (18.6) | 2066 (28.6)
Statistical Analysis 1: Comparison: Cohort 2: DOVATO (DTG/3TC) Fed vs Cohort 2: DOVATO (DTG/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.7284, 90% CI 2-sided [0.6576 to 0.8068] — An analysis of variance was performed on parameter Cmax for Analyte DTG to compare treatment arms Cohort 2: DOVATO (DTG/3TC) Fed with Cohort 2: DOVATO (DTG/3TC) Fasted
Statistical Analysis 2: Comparison: Cohort 2: DOVATO (DTG/3TC) Fed vs Cohort 2: DOVATO (DTG/3TC) Fasted; Test type: Other; Ratio of Geometric Least Square Means = 0.5191, 90% CI 2-sided [0.4535 to 0.5943] — An analysis of variance was performed on parameter Cmax for Analyte 3TC to compare treatment arms Cohort 2: DOVATO (DTG/3TC) Fed with Cohort 2: DOVATO (DTG/3TC) Fasted

7. Secondary Outcome: Cohort 1: Lag Time for Absorption (Tlag) of DTG, ABC and 3TC Following Administration of TRIUMEQ Under Fed and Fasted Conditions
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Hours
  DTG | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  ABC | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  3TC | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]

8. Secondary Outcome: Cohort 1: Terminal Elimination Phase Half-life (t1/2) of DTG, ABC and 3TC Following Administration of TRIUMEQ Under Fed and Fasted Conditions
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Hours
  DTG | 16.18 (21.0) | 16.10 (18.3)
  ABC | 2.291 (23.9) | 1.958 (28.4)
  3TC: number analyzed (Participants) | 15 | 16
  3TC | 17.35 (43.3) | 15.23 (52.9)

9. Secondary Outcome: Cohort 1: AUC From Time Zero to 24 Hours (AUC[0-24]) of DTG, ABC and 3TC Following Administration of TRIUMEQ Under Fed and Fasted Conditions
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12 and 24 Hours post dose in each treatment periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Hours*nanogram per milliliter
  DTG | 36380 (19.4) | 43870 (20.1)
  ABC | 8553 (24.8) | 9980 (28.8)
  3TC | 5817 (18.1) | 6707 (24.4)

10. Secondary Outcome: Cohort 1: Last Quantifiable Concentration (Ct) of DTG, ABC and 3TC Following Administration of TRIUMEQ Under Fed and Fasted Conditions
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Nanogram per milliliter
  DTG | 122.2 (69.6) | 128.6 (60.6)
  ABC | 10.61 (164.7) | 17.51 (124.9)
  3TC | 5.280 (32.3) | 4.621 (20.3)

11. Secondary Outcome: Cohort 1: Concentration at 24 Hours Post-dose (C24) of DTG, ABC and 3TC Following Administration of TRIUMEQ Under Fed and Fasted Conditions
Description: as for outcome 2
Time Frame: 24 hours post dose in treatment periods 1 and 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Nanogram per milliliter
  DTG | 958.6 (28.3) | 996.3 (26.3)
  ABC: number analyzed (Participants) | 10 | 4
  ABC | 4.833 (52.3) | 3.814 (27.2)
  3TC | 23.40 (24.4) | 21.74 (23.1)

12. Secondary Outcome: Cohort 1: Time of Maximum Observed Concentration (Tmax) of DTG, ABC and 3TC Following Administration of TRIUMEQ Under Fed and Fasted Conditions
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Hours
  DTG | 5.000 [3.00 to 12.00] | 1.250 [0.50 to 4.00]
  ABC | 2.750 [0.50 to 4.00] | 0.500 [0.25 to 1.50]
  3TC | 3.500 [2.00 to 4.00] | 1.508 [0.50 to 3.50]

13. Secondary Outcome: Cohort 2: Tlag of DTG and 3TC Following Administration of DOVATO Under Fed and Fasted Conditions
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 17 | 16
Hours
  DTG | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  3TC | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]

14. Secondary Outcome: Cohort 2: t1/2 of DTG and 3TC Following Administration of DOVATO Under Fed and Fasted Conditions
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Hours
  DTG | 14.43 (17.5) | 15.12 (19.0)
  3TC | 18.47 (28.8) | 18.36 (21.0)

15. Secondary Outcome: Cohort 2: AUC(0-24) of DTG and 3TC Following Administration of DOVATO Under Fed and Fasted Conditions
Description: as for outcome 4
Time Frame: as for outcome 9
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 17 | 16
Hours*nanogram per milliliter
  DTG | 32620 (19.2) | 35360 (15.6)
  3TC | 6339 (10.7) | 7339 (14.9)

16. Secondary Outcome: Cohort 2: Ct of DTG and 3TC Following Administration of DOVATO Under Fed and Fasted Conditions
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16
Nanogram per milliliter
  DTG | 82.37 (59.6) | 79.73 (74.5)
  3TC | 4.078 (29.6) | 3.622 (25.4)

17. Secondary Outcome: Cohort 2: C24 of DTG and 3TC Following Administration of DOVATO Under Fed and Fasted Conditions
Description: as for outcome 4
Time Frame: 24 hours post dose in treatment periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 17 | 16
Nanogram per milliliter
  DTG | 764.7 (28.5) | 715.4 (27.7)
  3TC | 22.56 (18.8) | 20.38 (18.6)

18. Secondary Outcome: Cohort 2: Tmax of DTG and 3TC Following Administration of DOVATO Under Fed and Fasted Conditions
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 17 | 16
Hours
  DTG | 4.000 [3.50 to 8.00] | 0.875 [0.50 to 3.50]
  3TC | 3.000 [0.75 to 4.00] | 0.750 [0.50 to 1.00]

19. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or other situations as per Medical or scientific judgment.
Time Frame: Up to 23 days
Population: Safety Population consisted of all participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Participants
  AEs | 1 | 3 | 1 | 1
  SAEs | 0 | 0 | 0 | 0

20. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count and Neutrophil
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils and platelet count. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
10^9 cells per liter
  Basophils | -0.002 (0.0105) | -0.004 (0.0141) | -0.003 (0.0100) | 0.001 (0.0144)
  Eosinophils | -0.002 (0.0456) | 0.015 (0.0755) | -0.005 (0.0219) | 0.006 (0.0318)
  Lymphocytes | -0.212 (0.3773) | -0.116 (0.2271) | -0.027 (0.2865) | -0.066 (0.3669)
  Monocytes | -0.051 (0.0972) | -0.048 (0.0802) | -0.064 (0.1285) | -0.021 (0.1169)
  Platelet count | 3.2 (16.05) | 6.7 (15.40) | 5.4 (23.00) | 5.5 (19.96)
  Neutrophil | 0.031 (0.5042) | -0.159 (0.6044) | -0.109 (0.9421) | -0.133 (0.9317)

21. Secondary Outcome: Change From Baseline in Hematology Parameters: Red Blood Cell (RBC) Count
Description: Blood samples were collected to analyze the hematology parameter: RBC count. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
10^12 cells per liter | 0.008 (0.1891) | -0.006 (0.1832) | 0.024 (0.2141) | 0.018 (0.1620)

22. Secondary Outcome: Change From Baseline in Hematology Parameters: Hemoglobin
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
Grams per liter | 0.3 (5.66) | -1.1 (4.96) | 1.2 (6.40) | -0.1 (5.17)

23. Secondary Outcome: Change From Baseline in Hematology Parameters: Hematocrit
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the hematology parameter: hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
Proportion of red blood cells in blood | -0.0001 (0.01647) | 0.0003 (0.01587) | 0.0006 (0.01950) | 0.0010 (0.01487)

24. Secondary Outcome: Change From Baseline in Hematology Parameters: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the hematology parameter: erythrocytes mean corpuscular Volume. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
Femtoliter | -0.09 (0.665) | 0.12 (0.571) | -0.28 (0.471) | -0.14 (0.672)

25. Secondary Outcome: Change From Baseline in Hematology Parameters: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
Picograms | -0.03 (0.267) | -0.24 (0.307) | 0.13 (0.442) | -0.09 (0.351)

26. Secondary Outcome: Absolute Values of Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count and Neutrophil
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils and platelet count. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
10^9 cells per liter
  Baseline (Day -1): Basophils | 0.040 (0.0210) | 0.043 (0.0202) | 0.042 (0.0144) | 0.041 (0.0200)
  Day 4: Basophils: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Basophils | 0.038 (0.0223) | 0.039 (0.0169) | 0.039 (0.0131) | 0.042 (0.0176)
  Baseline (Day -1): Eosinophils | 0.192 (0.0821) | 0.190 (0.1081) | 0.147 (0.0956) | 0.150 (0.0922)
  Day 4: Eosinophils: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Eosinophils | 0.190 (0.0989) | 0.205 (0.1231) | 0.144 (0.1022) | 0.156 (0.1050)
  Baseline (Day -1): Lymphocytes | 2.002 (0.5419) | 1.908 (0.4189) | 2.029 (0.5486) | 2.008 (0.5350)
  Day 4: Lymphocytes: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Lymphocytes | 1.790 (0.3956) | 1.793 (0.3677) | 1.922 (0.5003) | 1.941 (0.5713)
  Baseline (Day -1): Monocytes | 0.461 (0.2078) | 0.449 (0.1554) | 0.507 (0.1661) | 0.469 (0.1018)
  Day 4: Monocytes: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Monocytes | 0.409 (0.1335) | 0.402 (0.1373) | 0.435 (0.1185) | 0.448 (0.1222)
  Baseline (Day -1): Platelet count | 272.4 (66.59) | 276.8 (69.88) | 253.9 (56.34) | 243.1 (54.54)
  Day 4: Platelet count: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Platelet count | 275.6 (65.27) | 283.5 (64.14) | 249.8 (42.35) | 248.6 (55.33)
  Baseline (Day -1): Neutrophil | 3.299 (1.2456) | 3.407 (1.1862) | 3.436 (1.3351) | 3.436 (1.0628)
  Day 4: Neutrophil: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Neutrophil | 3.329 (0.9590) | 3.248 (0.8036) | 3.275 (1.4198) | 3.304 (1.5065)

27. Secondary Outcome: Absolute Values of Hematology Parameters: RBC Count
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the hematology parameters: RBC count. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
10^12 cells per liter
  Baseline (Day -1) | 4.648 (0.4082) | 4.684 (0.3549) | 4.765 (0.4251) | 4.848 (0.3975)
  Day 4: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4 | 4.656 (0.4170) | 4.678 (0.4011) | 4.839 (0.4405) | 4.865 (0.4051)

28. Secondary Outcome: Absolute Values of Hematology Parameters: Hemoglobin
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Grams per liter
  Baseline (Day -1) | 133.5 (16.66) | 134.4 (15.71) | 142.0 (11.69) | 144.5 (11.25)
  Day 4: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4 | 133.8 (16.66) | 133.3 (16.97) | 144.3 (12.06) | 144.4 (10.57)

29. Secondary Outcome: Absolute Values of Hematology Parameters: Hematocrit
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the hematology parameter: hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Proportion of red blood cells in blood
  Baseline (Day -1) | 0.3957 (0.04371) | 0.3976 (0.03892) | 0.4163 (0.03383) | 0.4227 (0.03075)
  Day 4: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4 | 0.3956 (0.04208) | 0.3979 (0.04358) | 0.4201 (0.03339) | 0.4237 (0.03137)

30. Secondary Outcome: Absolute Values of Hematology Parameters: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the hematology parameter: erythrocytes mean corpuscular Volume. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Femtoliter
  Baseline (Day -1) | 85.11 (5.706) | 84.92 (5.749) | 87.64 (5.684) | 87.45 (5.795)
  Day 4: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4 | 85.02 (5.470) | 85.04 (5.712) | 87.09 (5.648) | 87.31 (5.612)

31. Secondary Outcome: Absolute Values of Hematology Parameters: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Picograms
  Baseline (Day -1) | 28.74 (2.549) | 28.71 (2.655) | 29.89 (2.246) | 29.89 (2.210)
  Day 4: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4 | 28.71 (2.544) | 28.48 (2.592) | 29.92 (2.260) | 29.80 (2.241)

32. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP) and Aspartate Amino Transferase (AST)
Description: Blood samples were collected to analyze the clinical chemistry parameters: ALT, ALP and AST. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
International units per liter
  ALT | 4.0 (12.63) | -5.1 (7.02) | -0.4 (4.10) | -3.6 (5.06)
  ALP | -2.6 (5.71) | -3.0 (6.80) | 0.3 (4.51) | -1.6 (4.15)
  AST | 0.6 (6.69) | -4.0 (4.59) | -1.3 (1.70) | -2.0 (3.44)

33. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Calcium, Glucose, Potassium, Sodium and Blood Urea Nitrogen (BUN)
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the clinical chemistry parameters: calcium, glucose, potassium, sodium and BUN. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
Millimoles per liter
  Calcium | -0.003 (0.0436) | -0.034 (0.0781) | 0.029 (0.0792) | 0.038 (0.0674)
  Glucose | -0.037 (0.2700) | -0.169 (0.3648) | -0.047 (0.2156) | -0.049 (0.4082)
  Potassium | 0.03 (0.244) | 0.01 (0.189) | -0.13 (0.277) | -0.08 (0.434)
  Sodium | 0.4 (1.36) | 0.9 (1.29) | -0.5 (1.41) | 0.3 (1.40)
  BUN | 0.208 (0.4826) | 0.293 (0.8664) | 0.353 (0.8394) | 0.445 (0.9233)

34. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Creatinine, Direct Bilirubin and Total Bilirubin
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the clinical chemistry parameters: creatinine, direct bilirubin and total bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
Micromoles per liter
  Creatinine | 9.18 (2.871) | 10.76 (4.045) | 1.83 (2.931) | 2.11 (5.796)
  Direct Bilirubin | 0.16 (0.541) | 0.05 (0.398) | 0.04 (0.403) | -0.06 (0.330)
  Total Bilirubin | 0.16 (3.069) | -0.74 (2.712) | 0.58 (2.377) | -0.03 (1.588)

35. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Creatine Kinase
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the clinical chemistry parameters: creatine kinase. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
International units per liter | -17.8 (47.62) | -51.9 (82.52) | -33.9 (44.83) | -29.5 (91.10)

36. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Albumin and Total Protein
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the clinical chemistry parameters: albumin and total protein. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
Grams per liter
  Albumin | 0.2 (2.32) | -0.9 (3.20) | 0.9 (2.55) | 1.1 (1.67)
  Total Protein | 0.9 (3.07) | -0.2 (4.59) | 0.8 (3.58) | 0.7 (3.32)

37. Secondary Outcome: Absolute Values of Clinical Chemistry Parameters: ALT, ALP and AST
Description: Blood samples were collected to analyze the clinical chemistry parameters: ALT, ALP and AST. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
International units per liter
  Baseline (Day -1): ALT | 19.7 (9.16) | 24.3 (15.10) | 23.4 (16.38) | 24.8 (15.45)
  Day 4: ALT: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: ALT | 23.7 (18.71) | 19.3 (9.69) | 22.6 (16.01) | 21.1 (14.24)
  Baseline (Day -1) ALP | 66.8 (15.23) | 65.6 (17.65) | 59.3 (13.58) | 61.8 (14.65)
  Day 4: ALP: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: ALP | 64.1 (16.18) | 62.6 (14.47) | 60.1 (13.85) | 60.2 (13.16)
  Baseline (Day -1): AST | 18.4 (5.26) | 20.6 (5.77) | 18.5 (6.97) | 18.9 (6.57)
  Day 4: AST: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: AST | 19.0 (8.82) | 16.6 (2.94) | 17.3 (6.04) | 16.9 (5.11)

38. Secondary Outcome: Absolute Values of Clinical Chemistry Parameters: Calcium, Glucose, Potassium, Sodium and BUN
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the clinical chemistry parameters: calcium, glucose, potassium, sodium and BUN. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Millimoles per liter
  Baseline (Day -1): Calcium | 2.350 (0.1030) | 2.376 (0.0975) | 2.339 (0.0793) | 2.333 (0.0981)
  Day 4: Calcium: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Calcium | 2.347 (0.0899) | 2.342 (0.0980) | 2.368 (0.0742) | 2.371 (0.0721)
  Baseline (Day -1): Glucose | 4.821 (0.3214) | 5.016 (0.3793) | 4.974 (0.3943) | 5.068 (0.4760)
  Day 4: Glucose: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Glucose | 4.784 (0.2407) | 4.848 (0.2820) | 4.943 (0.4349) | 5.019 (0.3243)
  Baseline (Day -1): Potassium | 4.11 (0.268) | 4.16 (0.239) | 4.33 (0.335) | 4.31 (0.330)
  Day 4: Potassium: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Potassium | 4.14 (0.216) | 4.18 (0.224) | 4.23 (0.235) | 4.23 (0.298)
  Baseline (Day -1): Sodium | 137.8 (0.91) | 137.9 (1.67) | 138.5 (1.59) | 138.8 (1.73)
  Day 4: Sodium: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Sodium | 138.3 (1.73) | 138.8 (1.17) | 138.2 (1.47) | 139.1 (1.61)
  Baseline (Day -1): BUN | 4.531 (0.9081) | 4.333 (1.0302) | 4.633 (0.9609) | 4.592 (1.3875)
  Day 4: BUN: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: BUN | 4.739 (0.7250) | 4.626 (0.8416) | 5.065 (1.0791) | 5.037 (1.0406)

39. Secondary Outcome: Absolute Values of Clinical Chemistry Parameters: Creatinine, Direct Bilirubin and Total Bilirubin
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the clinical chemistry parameters: creatinine, direct bilirubin and total bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Micromoles per liter
  Baseline (Day -1): Creatinine | 74.38 (14.598) | 75.10 (15.407) | 80.18 (12.794) | 82.54 (9.056)
  Day 4: Creatinine: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Creatinine | 83.55 (15.394) | 85.86 (16.173) | 83.87 (10.444) | 84.65 (10.814)
  Baseline (Day -1): Direct Bilirubin | 1.88 (0.886) | 1.88 (0.748) | 1.74 (0.271) | 1.84 (0.505)
  Day 4: Direct Bilirubin: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Direct Bilirubin | 2.04 (0.776) | 1.93 (0.767) | 1.80 (0.539) | 1.78 (0.437)
  Baseline (Day -1): Total Bilirubin | 10.33 (4.305) | 10.63 (4.326) | 9.90 (2.286) | 10.55 (3.109)
  Day 4: Total Bilirubin: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Total Bilirubin | 10.49 (3.560) | 9.89 (3.747) | 10.73 (3.405) | 10.52 (3.040)

40. Secondary Outcome: Absolute Values of Clinical Chemistry Parameters: Creatine Kinase
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the clinical chemistry parameters: creatine kinase. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
International units per liter
  Baseline (Day -1) | 111.5 (66.68) | 143.8 (110.57) | 119.7 (59.78) | 124.6 (117.54)
  Day 4: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4 | 93.7 (47.08) | 91.8 (53.25) | 86.6 (34.64) | 95.1 (44.21)

41. Secondary Outcome: Absolute Values of Clinical Chemistry Parameters: Albumin and Total Protein
Description: Blood samples were collected at Baseline and at Day 4 post dose of each period to analyze the clinical chemistry parameters: albumin and total protein. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Grams per liter
  Baseline (Day -1): Albumin | 44.0 (3.31) | 44.5 (3.58) | 43.0 (2.57) | 42.9 (2.59)
  Day 4: Albumin: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Albumin | 44.2 (2.81) | 43.6 (2.83) | 43.7 (2.63) | 44.1 (2.86)
  Baseline (Day -1): Total Protein | 71.3 (3.82) | 71.8 (3.64) | 69.1 (4.32) | 69.4 (4.36)
  Day 4: Total Protein: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Total Protein | 72.2 (3.04) | 71.6 (2.90) | 69.6 (4.08) | 70.1 (4.91)

42. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected at Baseline and at Day 4 post dose of each period to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
Ratio | 0.0034 (0.00650) | 0.0013 (0.01116) | 0.0029 (0.00809) | 0.0019 (0.00570)

43. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Potential of Hydrogen (pH) by Dipstick
Description: Urine samples were collected at Baseline and at Day 4 post dose of each period to analyze the urinalysis parameter: pH by dipstick. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
pH | -0.34 (0.724) | -0.22 (0.547) | -0.13 (0.645) | -0.44 (0.512)

44. Secondary Outcome: Absolute Values of Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected at Baseline and at Day 4 post dose of each period to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Ratio
  Baseline (Day -1) | 1.0128 (0.00767) | 1.0134 (0.00766) | 1.0151 (0.00800) | 1.0163 (0.00857)
  Day 4: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4 | 1.0162 (0.00782) | 1.0147 (0.00921) | 1.0182 (0.00727) | 1.0181 (0.00851)

45. Secondary Outcome: Absolute Values of Urinalysis Parameter: Potential of Hydrogen (pH) by Dipstick
Description: Urine samples were collected at Baseline and at Day 4 post dose of each period to analyze the urinalysis parameter: pH by dipstick. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
pH
  Baseline (Day -1) | 6.38 (0.806) | 6.22 (0.515) | 6.41 (0.643) | 6.50 (0.548)
  Day 4: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4 | 6.03 (0.499) | 6.00 (0.577) | 6.28 (0.605) | 6.06 (0.544)

46. Secondary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick
Description: Urine samples were collected at indicated time points to analyze parameters including glucose, protein, blood, and ketones by dipstick. The dipstick test gives results in a semi-quantitative manner and results for urinalysis parameters can be read as Negative, Trace, 1+ (low concentrations present), 2+ (moderate concentrations present), 3+ (high concentrations present) and 4+ (very high concentrations present) indicating proportional concentrations in the urine sample.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Participants
  Baseline (Day -1): Urine Glucose (Negative) | 16 | 16 | 17 | 16
  Day 4: Urine Glucose (Negative): number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Urine Glucose (Negative) | 16 | 16 | 16 | 16
  Baseline (Day -1): Urine Protein (Negative) | 16 | 16 | 17 | 16
  Day 4: Urine Protein (Negative): number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Urine Protein (Negative) | 16 | 16 | 16 | 16
  Baseline (Day -1): Urine Blood (Negative) | 16 | 15 | 16 | 15
  Baseline (Day -1): Urine Blood (3+) | 0 | 1 | 0 | 0
  Baseline (Day -1): Urine Blood (2+) | 0 | 0 | 0 | 1
  Baseline (Day -1): Urine Blood (Trace) | 0 | 0 | 1 | 0
  Day 4: Urine Blood (Negative): number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Urine Blood (Negative) | 15 | 14 | 16 | 15
  Day 4: Urine Blood (2+): number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Urine Blood (2+) | 1 | 2 | 0 | 0
  Day 4: Urine Blood (3+): number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Urine Blood (3+) | 0 | 0 | 0 | 1
  Baseline (Day -1): Urine Ketones (Negative) | 16 | 16 | 17 | 16
  Day 4: Urine Ketones (Negative): number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Urine Ketones (Negative) | 15 | 16 | 16 | 16
  Day 4: Urine Ketones (1+): number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: Urine Ketones (1+) | 1 | 0 | 0 | 0

47. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters: PR Interval, QRS Duration, QT Interval and Corrected QT Interval According to Fridericia's Formula (QTcF)
Description: Single 12-lead ECGs were obtained to measure PR Interval, QRS Duration, QT Interval and QTcF Interval. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
Milliseconds
  PR Interval | 2.2 (9.70) | -0.7 (12.39) | -2.7 (9.90) | 4.0 (5.69)
  QRS Duration | -1.2 (3.35) | -2.9 (4.44) | 1.2 (2.99) | 0.1 (3.23)
  QT Interval | -10.5 (15.80) | -6.4 (17.20) | -13.1 (11.26) | -2.4 (13.86)
  QTcF | -4.1 (11.87) | -6.9 (11.21) | -2.5 (8.71) | -0.8 (6.10)

48. Secondary Outcome: Absolute Values of ECG Parameters: PR Interval, QRS Duration, QT Interval and QTcF
Description: Single 12-lead ECGs were obtained to measure PR Interval, QRS Duration, QT Interval and QTcF Interval. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Milliseconds
  Baseline (Day -1): PR Interval | 163.4 (24.29) | 161.6 (23.91) | 174.6 (25.55) | 176.1 (21.82)
  Day 4: PR Interval: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: PR Interval | 165.6 (23.35) | 160.9 (24.82) | 174.8 (17.72) | 180.1 (19.48)
  Baseline (Day -1): QRS Duration | 95.6 (8.66) | 96.7 (10.62) | 93.4 (8.12) | 93.1 (7.27)
  Day 4: QRS Duration: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: QRS Duration | 94.4 (8.38) | 93.8 (10.36) | 93.8 (7.48) | 93.2 (7.53)
  Baseline (Day -1): QT Interval | 401.8 (21.90) | 400.7 (21.35) | 407.5 (23.85) | 402.2 (25.69)
  Day 4: QT Interval: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: QT Interval | 391.3 (15.10) | 394.3 (19.00) | 392.9 (20.51) | 399.8 (25.41)
  Baseline (Day -1) | 400.1 (14.30) | 403.6 (14.51) | 400.1 (17.84) | 401.3 (16.99)
  Day 4: QTcF: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: QTcF | 395.9 (14.26) | 396.6 (13.34) | 395.6 (19.23) | 400.4 (18.54)

49. Secondary Outcome: Change From Baseline in Vital Signs Measurements: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in the supine or semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
Millimeters of mercury
  SBP | -1.1 (4.32) | -4.2 (6.71) | 1.9 (8.14) | 0.6 (8.54)
  DBP | 0.0 (7.27) | 0.3 (5.20) | 3.0 (6.46) | -1.1 (8.71)

50. Secondary Outcome: Absolute Values of Vital Signs Measurements: SBP and DBP
Description: SBP and DBP were measured in the supine or semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Millimeters of mercury
  Baseline (Day -1): SBP | 110.6 (10.61) | 113.0 (10.04) | 112.5 (9.37) | 113.5 (8.65)
  Day 4: SBP: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: SBP | 109.5 (10.93) | 108.8 (9.07) | 114.7 (9.14) | 114.1 (10.67)
  Baseline (Day -1): DBP | 64.0 (7.68) | 64.0 (7.69) | 63.0 (7.37) | 66.4 (6.55)
  Day 4: DBP: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4: DBP | 64.0 (9.12) | 64.3 (8.99) | 66.4 (8.06) | 65.3 (8.20)

51. Secondary Outcome: Change From Baseline in Vital Signs Measurements: Pulse Rate
Description: Pulse rate were measured in the supine or semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 16
Beats per minute | 3.0 (5.18) | -0.3 (5.87) | 1.1 (10.12) | -0.1 (7.04)

52. Secondary Outcome: Absolute Values of Vital Signs Measurements: Pulse Rate
Description: Pulse rate were measured in the supine or semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
Number analyzed (Participants) | 16 | 16 | 17 | 16
Beats per minute
  Baseline (Day -1) | 59.9 (9.07) | 62.3 (7.49) | 59.9 (10.82) | 60.1 (8.44)
  Day 4: number analyzed (Participants) | 16 | 16 | 16 | 16
  Day 4 | 62.9 (8.47) | 62.0 (9.89) | 61.4 (3.86) | 59.9 (6.68)

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious Adverse Events (SAEs) and non-SAEs were collected up to 23 days.
Description: All-cause mortality, SAEs and non-SAEs were reported for Safety Population that consisted of all participants who received at least one dose of study intervention. Adverse events were presented treatment-wise.
Arm/Group | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted | Cohort 2: DOVATO (DTG/3TC) Fed | Cohort 2: DOVATO (DTG/3TC) Fasted
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 3/16 | 1/17 | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fed (N=16) | Cohort 1: TRIUMEQ (DTG/ABC/3TC) Fasted (N=16) | Cohort 2: DOVATO (DTG/3TC) Fed (N=17) | Cohort 2: DOVATO (DTG/3TC) Fasted (N=16)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT04827134/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT04827134/SAP_001.pdf